CLINICAL TRIAL: NCT02565394
Title: OR-STRETCH: Microbreaks in the Operating Room With the Incorporation of Stretches to Mitigate High Physical and Mental Demands While Enhancing Performance During Surgical Procedures
Brief Title: Microbreaks in the OR to Mitigate High Physical and Mental Demands
Acronym: OR-STRETCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Susan Hallbeck, Ph.D., Senior Associate Consultant II, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-006129
Record Dates: First submitted 2015-08-13; First posted 2015-10-01 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Attention Concentration Difficulty; Neck Pain; Back Pain; Shoulder Pain; Fatigue
MeSH Terms: conditions — Neck Pain; Back Pain; Shoulder Pain; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micro-Break with Dynamic Activity (Experimental): Micro Break with web based application of a video to lead surgeons through dynamic exercise activities
  Interventions: Other: Micro Break with Dynamic Exercise Activities
- Comparator (No Intervention): A baseline survey will be completed following a surgical day with no dynamic activities

INTERVENTIONS:
Other: Micro Break with Dynamic Exercise Activities — Surgeons may elect to activate a web application (video) and perform targeted intraoperative exercises.
  Arms: Micro-Break with Dynamic Activity

SUMMARY:
Will targeted intraoperative exercises performed by surgeons during surgery, mitigate high physical and mental demands while enhancing performance during surgical procedures?

DETAILED DESCRIPTION:
This study will compare the efficacy of incorporating dynamic exercises into the surgical procedure, to determine if the exercise intervention will decrease surgeon's perceived physical discomfort and fatigue and enhance self-reported performance during surgical procedures. All attending surgeons (Cardiothoracic, Colon and Rectal, General, Gynecology and Obstetrics, Ophthalmic, Orthopedic, Otolaryngology-Head and Neck, Neurology, Urology, Plastic and Maxillofacial, Rural, Urology, Thoracic and Vascular ) or surgeons in training that are board certified or board eligible, performing open or minimally invasive surgery within the scope of their practice in the house of surgery at Mayo Clinic Rochester, Arizona and Florida will be eligible to participate. Surgeons who have provided informed consent to participate will be asked to complete a preliminary baseline survey that will provide information regarding baseline participant characteristics and demographics.

The intervention is a web based application which will include a short video with verbal cues, available on computers in the Operating Rooms (ORs). This video will lead surgeons through the stretch exercises and include a timer to remind them when it is time to stretch. They will be able to set the time interval between stretches (between 20-55 minutes) and may activate a snooze on the timer to postpone the stretch to a more opportune time during the procedure. The stretches can be performed without breaking scrub, in the sterile field and can be completed in approximately 1 minute.

Surgeons will be asked to participate in this study for approximately 12 weeks , completing a baseline survey and three end of day surveys. They may use the intervention as much or as little as they choose during their participation, and will be free to use the application following study participation. The web application does track participant use, providing date and time stamps to enable the research team to track surgeon web app utilization. The application will also record how often the "snooze" was used to delay a stretch, or end stretches. After surgeons have accessed the web application, they will receive an email with a quick survey about their experiences with stretches, to assess the impact of the web app.

ELIGIBILITY:
Inclusion Criteria:

1. Attending surgeons (Cardiothoracic, Colon and Rectal, General, Gynecology and Obstetrics, Ophthalmic, Orthopedic, Otolaryngology-Head and Neck, Neurology, Urology, Plastic and Maxillofacial, Rural, Urology, Thoracic and Vascular ) or surgeons in training that are board certified or board eligible, performing open or minimally invasive surgery within the scope of their practice in the house of surgery at Mayo Clinic Rochester
2. Over the age of 21
3. As feasible, equal numbers of males, females and minorities
4. Performing greater than 50% of the surgery

Exclusion Criteria:

1. Participants who are visibly unwell or report being unwell at time of study
2. Participants unable to devote the minimum time required to complete study procedures

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Decrease in surgeon's perceived physical discomfort and fatigue following surgeries where the dynamic exercises were performed as measured by questionnaire | baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hallbeck, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota